CLINICAL TRIAL: NCT02464878
Title: Multicenter Trial of the Effect of AAT on Islet Transplant Engraftment and Durability After Renal Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Iowa (Other)
Responsible Party: Principal Investigator, James F. Markmann, MD, PhD, Chief, Division of Transplant Surgery, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Islet after Kidney - AAT
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Results first posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-11

CONDITIONS: Kidney Transplant; Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — alpha 1-Antitrypsin; Islets of Langerhans Transplantation; thymoglobulin; Antilymphocyte Serum; Basiliximab; Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- Main study treatment (Other)
  Interventions: Drug: Alpha 1-Antitrypsin; Procedure: Islet Transplantation; Drug: Thymoglobulin; Drug: Basiliximab; Drug: Etanercept

INTERVENTIONS:
Drug: Alpha 1-Antitrypsin — Patients will receive three times a week AAT infusions in the peri-transplant period for three weeks.
  Other Names: Glassia
Procedure: Islet Transplantation
Drug: Thymoglobulin — Patients will receive a total of 5 doses between Day -2 and Day +2
  Other Names: Antithymocyte Globulin
Drug: Basiliximab — Basiliximab will be used for subsequent transplants.
Drug: Etanercept — Etanercept will be given on the day of transplant and on Days 3, 7, and 10 post-transplant.
  Other Names: Enbrel

SUMMARY:
Patients meeting the study entry criteria will receive 1-3 infusion(s) of in vitro cultured islets. Patients will receive three times a week AAT infusions in the peri-transplant period for three weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects age 18 to 70 years.
* Subjects who are able to provide written informed consent and to comply with the procedures of the study protocol.
* Subjects must have one of the following payment mechanisms in place:

  1. Medicare,
  2. A third-party insurer who agrees, via pre-authorization, to pay for participation in the study, or
  3. Another mechanism of payment (self-pay, hospital, university, donations, etc.) for participation in the study.
* Clinical history compatible with T1D with disease onset < 40 years of age and insulin-dependence for ≥ 5 years at the time of enrollment.
* Absent stimulated c-peptide (< 0.3 ng/mL) in response to a MMTT [Boost® 6 mL/kg body weight (BW) to a maximum of 360 mL; another product with equivalent caloric and nutrient content may be substituted for Boost®] measured at 60 and 90 min after start of consumption.
* Subjects who are ≥ 3 months post-renal transplant who are taking appropriate calcineurin inhibitor (CNI) based maintenance immunosuppression ([tacrolimus alone or in conjunction with sirolimus, mycophenolate mofetil, myfortic, or azathioprine; or cyclosporine in conjunction with sirolimus, mycophenolate mofetil, or myfortic] ± Prednisone ≤ 10 mg/day).
* Stable renal function as defined by a creatinine of no more than one third greater than the average creatinine determination performed in the 3 previous months prior to islet transplantation, until rejection, obstruction or infection is ruled out.
* Subjects who meet one of the options in the following criterion are eligible for transplantation:

  * Reduced awareness of hypoglycemia manifested by a Clarke score of 4 or more measured upon study enrollment and at least one episode of severe hypoglycemia in the 12 months prior to study enrollment.
  * A subject must have a reduced awareness of hypoglycemia manifested by a Clarke score of 4 or more and at least 1 episode of severe hypoglycemia;
  * Any subject not meeting the hypoglycemia option must have an HbA1c > 7.5%.

Exclusion Criteria:

* Weight more than 100 kg or body mass index (BMI) > 33 kg/m2.
* Insulin requirement of >1.0 U/kg/day or, > 60 U/day total, or <15 U/day.
* Other (non-kidney) organ transplants except prior failed pancreatic graft where graft failure is attributed to thrombosis within the first 4 weeks or to other technical reasons that require graft pancreatectomy; with the graft pancreatectomy occurring more than 6 months ago.
* Untreated or unstable proliferative diabetic retinopathy.
* Blood Pressure: SBP > 160 mmHg or DBP >100 mmHg despite treatment with antihypertensive agents.
* Calculated GFR of ≤ 40 mL/min/1.73 m2 using the subject's measured serum creatinine and the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation1. Strict vegetarians (vegans) will be excluded only if their estimated GFR is ≤ 35 mL/min/1.73 m2.

  7. Proteinuria (albumin/creatinine ratio or ACr > 300mg/g) of new onset since kidney transplantation.
* Calculated panel-reactive anti-HLA antibodies > 50%. Subjects with calculated panel reactive anti-HLA antibodies ≤ 50% will be excluded if any of the following are detected:

  * Positive cross-match,
  * Islet donor-directed anti-HLA antibodies detected by Luminex Single Antigen/specificity bead assay including weakly reactive antibodies that would not be detected by a flow cross-match, or
  * Antibodies to the renal donor (i.e. presumed de novo).
* For female subjects: Positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of the study and 4 months after discontinuation. For male subjects: intent to procreate during the duration of the study or within 4 months after discontinuation or unwillingness to use effective measures of contraception. Oral contraceptives, Norplant®, Depo-Provera®, and barrier devices with spermicide are acceptable contraceptive methods; condoms used alone are not acceptable.
* Presence or history of active infection including hepatitis B, hepatitis C, HIV, or tuberculosis (TB). Subjects with laboratory evidence of active infection are excluded even in the absence of clinical evidence of active infection.
* Negative screen for Epstein-Barr virus (EBV) by IgG determination at time of screening or previous kidney transplant.
* Invasive aspergillus, histoplasmosis, and coccidoidomycosis infection within the last year.
* Any history of malignancy except for completely resected squamous or basal cell carcinoma of the skin.
* Known active alcohol or substance abuse.
* Any coagulopathy or medical condition requiring long-term anticoagulant therapy (e.g. warfarin) after islet transplantation (low-dose aspirin treatment [325 mg PO] is allowed) or subjects with international normalized ratio (INR) > 1.5. The use of Plavix is allowed only in conjunction with mini- laparotomy procedure at the time of islet transplant.
* Severe co-existing cardiac disease, characterized by any one of these conditions:

  * Recent MI (within past 6 months);
  * Evidence of ischemia on functional cardiac exam within the last year;
  * Left ventricular ejection fraction < 30%; or
  * Valvular disease requiring replacement with prosthetic valve.
* Persistent serum glutamic-oxaloacetic transaminase (SGOT [AST]), serum glutamate pyruvate transaminase (SGPT [ALT],) alkaline phosphatase or total bilirubin, with values > 1.5 times normal upper limits will exclude a subject.
* Active infections (except mild skin and nail fungal infections).
* Acute or chronic pancreatitis.
* Active peptic ulcer disease, symptomatic gallstones, or portal hypertension.
* Use of any investigational agents within 4 weeks of enrollment.
* Administration of live attenuated vaccine(s) within 2 months of enrollment.
* Any medical condition that, in the opinion of the investigator, will interfere with the safe participation in the trial. (Cancer screenings should be performed per current American Cancer Society guidelines).
* Positive screen for BK virus by polymerase chain reaction (PCR) performed at time of screening.
* A kidney transplant patient with type 1 diabetes who has an HbA1c < 7.5 and no history of severe hypoglycemia.
* Selective or severe IgA deficiency (levels < 5-7 mg/dL)
* AAT deficiency (defined as < 1.0ng/mg AAT)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2022-11 (Actual); Study Completion 2022-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Markmann, M.D. Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Main Study Treatment: Alpha 1-Antitrypsin: Patients will receive three times a week AAT infusions in the peri-transplant period for three weeks.
  Islet Transplantation
  Thymoglobulin: Patients will receive a total of 5 doses between Day -2 and Day +2
  Basiliximab: Basiliximab will be used for subsequent transplants.
  Etanercept: Etanercept will be given on the day of transplant and on Days 3, 7, and 10 post-transplant.
Period: Overall Study
Arm/Group | Main Study Treatment
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Main Study Treatment
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 51 [44 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of GLASSIA Versus Control CIT06 Subjects Achieving Insulin Independence After First Infusion of Single Donor Islets.
Description: Insulin Independence examined 75 days after 1st infusion; subject considered to be insulin independent if they are able to titrate off insulin therapy for <1 week AND all of the following are met:
  1. one HbA1c level, one fasting serum glucose level, and a Mixed Meal Tolerance Test (MMTT) documented within the visit window at Day 75 (Day 70-80) and 7 days of blood sugar and insulin readings are documented within +/- 7 days of the visit window (Day 63-87);
  2. HbA1c </= 6.5% or a >/= 2.5% decrease from baseline (within 91 days prior to transplant);
  3. fasting capillary glucose level should not exceed 140 mg/dL more than 3 times in 7 consecutive days;
  4. post-prandial serum glucose </= 180 mg/dL at 90 minutes during MMTT;
  5. fasting serum glucose level </= 126 mg/dL; (6) at least one MMTT fasting or stimulated c-peptide >/= 0.5 ng/mL
Time Frame: Day 75
Population: Due to reduced enrollment in study, unable to make statistically appropriate comparison between subjects receiving GLASSIA and Control CIT06 subjects from NCT00468117. Information provided is pertinent to the two subjects enrolled based on descriptions of Primary and Secondary Outcomes
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Treatment
Number analyzed (Participants) | 2
Participants
  Ability to titrate of insulin therapy for at least 1 week | 0
  Documented HbA1c, fasting serum glucose level, MMTT, & 7 days blood sugar/insulin readings | 2
  HbA1c ≤ 6.5% or a ≥ 2.5% decrease from baseline (within 91 days prior to transplant) | 2
  Fasting capillary glucose level should not exceed 140 mg/dL more than 3 x in 7 consecutive days | 1
  Post-prandial serum glucose ≤ 180 mg/dL at 90 minutes during the MMTT | 1
  Fasting serum glucose level ≤ 126 mg/dL | 1
  At least one MMTT fasting or stimulated c-peptide ≥ 0.5 ng/mL | 2

2. Secondary Outcome: The Proportion of GLASSIA Treated Versus Control CIT06 Subjects Who Are Insulin Independent After 1 or More Islet Infusions
Description: Subject considered to be insulin independent if they are able to titrate off insulin therapy for <1 week AND all of the following are met:
  1. one HbA1c level, one fasting serum glucose level, and a Mixed Meal Tolerance Test (MMTT) documented within the visit window of time frame, noted below, and 7 days of blood sugar and insulin readings are documented within +/- 7 days of the visit window;
  2. HbA1c </= 6.5% or a >/= 2.5% decrease from baseline (within 91 days prior to transplant);
  3. fasting capillary glucose level should not exceed 140 mg/dL more than 3 times in 7 consecutive days;
  4. post-prandial serum glucose </= 180 mg/dL at 90 minutes during MMTT;
  5. fasting serum glucose level </= 126 mg/dL;
  6. at least one MMTT fasting or stimulated c-peptide >/= 0.5 ng/mL
Time Frame: 1 year after the first islet infusion, 1 year after the last islet infusion, 2 years after the first islet infusion, 2 years after the last islet infusion
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Treatment
Number analyzed (Participants) | 2
Participants
  1 yr after 1st infusion | 2
  1 yr after last infusion | 1
  2 yrs after 1st infusion | 1
  2 yrs after last infusion | 1

3. Secondary Outcome: The Proportion of GLASSIA Treated Versus CIT06 Control Subjects With Both an HbA1c ≤ 6.5% AND an Absence of Severe Hypoglycemic Events
Description: Number of subjects with both an HbA1c </= 6.5% and no severe hypoglycemic events at specified timepoints; data utilized for measure were HbA1c levels and number of severe hypoglycemic events.
Time Frame: From Day 28 to Day 365 after the first islet transplant, From Day 28 to Day 730 after the first islet transplant.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Treatment
Number analyzed (Participants) | 2
Participants
  Day 28-365 after 1st infusion | 2
  Day 28-730 after 1st infusion | 1

4. Secondary Outcome: The Proportion of GLASSIA Treated Versus Control Subjects With Both an HbA1c < 7.0% AND Free of Severe Hypoglycemic Events
Description: Subjects with an HbA1c <7.0% and free of severe hypoglycemic events at specified timepoints; data utilized were HbA1c levels and number/absence of severe hypoglycemic events
Time Frame: From Day 28 to Day 365 after the first islet transplant, From Day 28 to Day 730 after the first islet transplant.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Treatment
Number analyzed (Participants) | 2
Participants
  Day 28-365 after 1st infusion | 2
  Day 28-730 after 1st infusion | 1

5. Secondary Outcome: The Proportion of GLASSIA Treated Versus Control CIT06 Subjects A Reduction in HbA1c of 1 Point AND an Absence of Severe Hypoglycemia
Description: Subjects with a reduction in HbA1c of 1 point and no severe hypoglycemia at specific timepoints. Data utilized were HbA1c numbers at specified timepoints and absence of any severe hypoglycemic events
Time Frame: From Day 28 to Day 365 after the first islet transplant, From Day 28 to Day 730 after the first islet transplant.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Treatment
Number analyzed (Participants) | 2
Participants
  Day 28-365 after 1st infusion | 1
  Day 28-730 after 1st infusion | 1

6. Secondary Outcome: The Change in Clarke Score From Baseline in GLASSIA Treated Versus Control CIT06 Subjects
Description: Clarke Score is a 7 question patient report of hypoglycemia awareness. Answers provide a rating of either A (aware) or R (reduced). Four or more R ratings suggest impaired hypoglycaemia awareness; < or equal to 2 = normal awareness, 3=borderline. A higher Clarke Score indicates reduced awarness.
Time Frame: 1 year and 2 years after the first islet transplant
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Treatment
Number analyzed (Participants) | 2
Participants
  Year 1 after 1st Infusion : Clarke Score improved from Baseline | 1
  Year 1 after 1st Infusion : Clarke Score without improvement from Baseline | 1
  Year 2 after 1st Infusion : Clarke Score improved from Baseline | 1
  Year 2 after 1st Infusion : Clarke Score without improvement from Baseline | 1

7. Secondary Outcome: The Proportion of Subjects Receiving a Second Islet Transplant Comparing GLASSIA Treated Versus Control CIT06 Subjects
Description: Subjects requiring a 2nd islet infusion at specified timepoints; data utilized were the number of patients who were not successful at gaining and maintaining insulin independence following the 1st infusion and required a 2nd infusion/transplant of islets.
Time Frame: 1 year and 2 years following the first and last islet transplant(s)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Treatment
Number analyzed (Participants) | 2
Participants
  1 yr after 1st infusion | 2
  1 yr after last infusion | 2
  2 yrs after 1st infusion | 2
  2 yrs after last infusion | 2

8. Secondary Outcome: The Proportion of Subjects Receiving a Third Islet Transplant Comparing GLASSIA Treated Versus Control CIT06 Subjects
Description: Number of subjects requiring a 3rd islet infusion. Data utilized were the number of patients require a 3rd transplant/infusion of islets due to continued requirement of insulin during study participation.
Time Frame: 1 year and 2 years following the first and last islet transplant(s)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Treatment
Number analyzed (Participants) | 2
Participants
  1 yr after 1st infusion | 0
  1 yr after last infusion | 0
  2 yrs after 1st infusion | 0
  2 yrs after last infusion | 0

9. Secondary Outcome: Cardiovascular Events [Death, Cerebrovascular Accident (CVA), Myocardial Infarction (MI)] and Changes in Atherogenic Profile for GLASSIA Treated Versus Control Subjects
Description: Subjects experience of cardiovascular events and changes in atherogenic profile were examined for the timepoints listed below. Data utilized were baseline lipid labs (triglycerides, total cholesterol, HDL, LDL, and Non-HDL Cholesterol) and lipid labs taken at specified timepoints. An improvement would be an overall improvement of the lipid profile (e.g. reduction in non-HDL cholesterol/overall cholesterol, decrease in LDL, increase in HDL, etc.). Due to the COVID-19 pandemic and increased risk faced by transplant/immunosuppressed individuals, some lipid labs were not collected and data has been indicated as NA due to reduction in sample collection/prioritizing safety labs for subjects.
Time Frame: 1 year and 2 years following the first and last islet transplant(s)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Treatment
Number analyzed (Participants) | 2
Participants
  1 yr after 1st infusion: Number of subjects experiencing a cardiovascular event | 0
  1 yr after 1st infusion: Subjects with improvement in Atherogenic Profile at timepoint compared to baseline | NA — Due to COVID-19 pandemic, some lipid labs were not done at required time point; data points are not available for either one or both subjects making outcome impossible to assess.
  1 yr after 1st infusion: Subjects with worsening Atherogenic Profile at timepoint compared to baseline | NA — Due to COVID-19 pandemic, some lipid labs were not done at required time point; data points are not available for either one or both subjects making outcome impossible to assess.
  1 yr after 1st infusion: Subjects without change to Atherogenic Profile at timepoint compared to baseline | NA — Due to COVID-19 pandemic, some lipid labs were not done at required time point; data points are not available for either one or both subjects making outcome impossible to assess.
  1 yr after last infusion: Number of subjects experiencing a cardiovascular event | 0
  1 yr after last infusion: Subjects with improvement in Atherogenic Profile at timepoint compared to baseline | 1
  1 yr after last infusion: Subjects with worsening Atherogenic Profile at timepoint compared to baseline | 0
  1 yr after last infusion: Subjects without change to Atherogenic Profile at timepoint compared to baseline | 1
  2 yrs after 1st infusion: Number of subjects experiencing a cardiovascular event | 0
  2 yrs after 1st infusion: Subjects with improvement in Atherogenic Profile at timepoint compared to baseline | NA — Due to COVID-19 pandemic, some lipid labs were not done at required time point; data points are not available for either one or both subjects making outcome impossible to assess.
  2 yrs after 1st infusion: Subjects with worsening Atherogenic Profile at timepoint compared to baseline | NA — Due to COVID-19 pandemic, some lipid labs were not done at required time point; data points are not available for either one or both subjects making outcome impossible to assess.
  2 yrs after 1st infusion: Subjects without change to Atherogenic Profile at timepoint compared to baseline | NA — Due to COVID-19 pandemic, some lipid labs were not done at required time point; data points are not available for either one or both subjects making outcome impossible to assess.
  2 yrs after last infusion: Number of subjects experiencing a cardiovascular event | 0
  2 yrs after last infusion: Subjects with improvement in Atherogenic Profile at timepoint compared to baseline | 0
  2 yrs after last infusion: Subjects with worsening Atherogenic Profile at timepoint compared to baseline | 0
  2 yrs after last infusion: Subjects without change to Atherogenic Profile at timepoint compared to baseline | 2

ADVERSE EVENTS:
Time Frame: 2 Years
Arm/Group | Main Study Treatment
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study Treatment (N=2)
Seizure (Nervous system disorders) | 1 (1)
Tounge Swelling (Allergic Reaction) (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study Treatment (N=2)
Abdominal Pain/Bloating (Gastrointestinal disorders) | 1 (2)
Chest Pain (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diaphoresis (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Elevated Creatinine (Infections and infestations) | 1 (1)
Elevated Liver Function Tests (Investigations) | 1 (1)
Fever (Investigations) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (4)
Shingles (Infections and infestations) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT02464878/Prot_SAP_000.pdf